CLINICAL TRIAL: NCT07327489
Title: Predicting Response to Immunotherapy From Analysis of Live Tumor Biopsies
Acronym: ELEPHAS-05
Status: Recruiting | Type: Observational
Sponsor: Elephas (Industry)
Responsible Party: Sponsor
Other Study IDs: ELEPHAS-05
Record Dates: First submitted 2025-12-19; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Immunotherapy; Advanced Solid Tumors Cancer; Bladder Cancer; TNBC, Triple Negative Breast Cancer; Colorectal Cancer; DMMR Colorectal Cancer; MSI-H Colorectal Cancer; Endometrial Cancer; Head and Neck Cancer; Kidney Cancer; Liver Cancer; NSCLC (Non-small-cell Lung Cancer); Skin Cancer; Melanoma (Skin Cancer)
Keywords: Immunotherapy; Live Tumor Biopsy; Elephas; Cancer; Imaging; Tumor Cutting; Treatment Response; Core Needle Biopsy; Forceps Biopsy; Punch Biopsy
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Liver Neoplasms; Carcinoma, Non-Small-Cell Lung; Skin Neoplasms; Melanoma | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Remaining specimens or specimen derivatives (e.g. H&E slides) may be banked indefinitely.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Adults aged 18 years or older, who are able and willing to provide written informed consent, have a suspected or confirmed cancer diagnosis and will be undergoing a biopsy or similar procedure to obtain tumor tissue as a normal course of their medical management or diagnostic work-up.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Subjects must be clinically able, at investigator discretion, to undergo additional biopsy passes during their biopsy. Biopsy specimen(s) will be obtained during a standard of care (SOC) procedure. If a subject receives a subsequent SOC biopsy for clinical diagnosis purposes, additional sample(s) may be collected and sent to the Sponsor.

SUMMARY:
This study will collect tumor specimens with correlated clinical and demographic data from patients who are undergoing a biopsy or similar procedure to obtain tumor tissue as a normal course of their medical management or diagnostic work-up for suspected or confirmed cancer.

DETAILED DESCRIPTION:
Elephas is researching mechanisms of cutting, sorting and imaging tumors that leave the 3D tumor microenvironment (TME), including its immune cells, intact. This allows qualitative and semi-quantitative identification and characterization of the ex vivo response to exposure of potential immunotherapy. The ex vivo response data will then be compared to the clinical real world response data to inform development efforts.

This study will collect tumor specimens from patients with suspected or confirmed cancer. These specimens, along with clinical data and genomic data obtained as part of a patient's standard of care, will be used to perform this research.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent for participation
2. Age ≥18 years at time of consent.
3. Have a suspected or confirmed cancer diagnosis that is to be evaluated by means of a biopsy.
4. Subjects who are newly diagnosed or have suspected cancer must be treatment-naïve at the time of biopsy. All other subjects should have the biopsy performed before starting their next line of treatment.

Exclusion Criteria:

1. Have a known auto-immune disease or prior condition (prior organ transplant, chronic kidney or liver disease) that renders them ineligible for immunotherapy (IO) treatment.
2. Severely immunocompromised person(s). Examples include patients on immunosuppressants, HIV positive patients on antiretrovirals, post transplantation patients.
3. Pregnant person(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older, who are able and willing to provide written informed consent, have a suspected or confirmed cancer diagnosis and will be undergoing a biopsy or similar procedure to obtain tumor tissue as a normal course of their medical management or diagnostic work-up.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2035-04 (Estimated); Study Completion 2038-04 (Estimated)

PRIMARY OUTCOMES:
Predicting In-Vivo Clinical Response to Immune Checkpoint Inhibitors & Researching Mechanisms of Tumor Cutting and Imaging | Study duration is approximately 36 months from enrollment to end of study.
  Collect human tumor specimens to research mechanisms of tumor cutting, imaging, and ex-vivo immunotherapy treatment response, while maintaining cell stability in a live tumor microenvironment.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Mercy Hospital - FTS, Fort Smith, Arkansas
  - Frederick Health Hospital, Frederick, Maryland
  - Mercy Hospital - SPG, Springfield, Missouri
  - Mercy Hospital - South, St Louis, Missouri
  - Mercy Hospital -STL, St Louis, Missouri
  - Mercy Hospital - OKC, Oklahoma City, Oklahoma
  - JPS Health Network, Forth Worth, Texas
  - Baylor Scott and White Biorepository, Temple, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen S, Zhang Z, Zheng X, Tao H, Zhang S, Ma J, Liu Z, Wang J, Qian Y, Cui P, Huang D, Huang Z, Wu Z, Hu Y. Response Efficacy of PD-1 and PD-L1 Inhibitors in Clinical Trials: A Systematic Review and Meta-Analysis. Front Oncol. 2021 Apr 16;11:562315. doi: 10.3389/fonc.2021.562315. eCollection 2021. PMID 33937012
- [Background] Cherukuri AR, Lubner MG, Zea R, Hinshaw JL, Lubner SJ, Matkowskyj KA, Foltz ML, Pickhardt PJ. Tissue sampling in the era of precision medicine: comparison of percutaneous biopsies performed for clinical trials or tumor genomics versus routine clinical care. Abdom Radiol (NY). 2019 Jun;44(6):2074-2080. doi: 10.1007/s00261-018-1702-1. PMID 30032384